CLINICAL TRIAL: NCT07235475
Title: Comparison Between the Analgesic Effect of Fascia Transversalis Block vs Caudal Block in Pediatrics Undergoing Inguinal Hernia Surgeries: Randomized Double-blinded Comparative Study
Brief Title: Comparison Between the Analgesic Effect of Fascia Transversalis Block vs Caudal Block
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, AbdElKhalik Mahmoud Shaban, Lecturer of anaesthesia, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MS-393-2025
Record Dates: First submitted 2025-11-14; First posted 2025-11-19 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Post Operative Pain, Acute
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fascia Transversalis Block (Active Comparator): Patients will receive Fascia Transversalis Block
  Interventions: Procedure: Fascia Transversalis Block
- caudal block (Active Comparator): Patients will receive caudal block
  Interventions: Procedure: Caudal Block Anesthesia

INTERVENTIONS:
Procedure: Caudal Block Anesthesia — Patients will receive a caudal block with 0.5 mL/kg of Bupivacaine 0.25% injected. The commercial preparation that will be used is Bupivacaine HCl (Sunny Pharmaceutical, Egypt)
  Arms: caudal block
Procedure: Fascia Transversalis Block — Patients will receive Fascia Transversalis Block using 0.5 mL/kg of Bupivacaine 0.25% . The commercial preparation that will be used is Bupivacaine HCl (Sunny Pharmaceutical, Egypt)
  Arms: Fascia Transversalis Block

SUMMARY:
Despite the growing interest in interfascial blocks and their successful use in pediatric surgeries, no previous randomized clinical trials have directly compared the analgesic efficacy, opioid-sparing effect, and safety profile of the fascia transversalis block versus the caudal block in pediatric patients undergoing unilateral inguinal hernia repair. This study aims to address this gap by providing the first head-to-head randomized comparison between both blocks in a standardized surgical setting

ELIGIBILITY:
Inclusion Criteria:

* ASA physical status I or II, scheduled for elective unilateral inguinal hernia surgery under general anesthesia

Exclusion Criteria:

* Parental refusal.
* Pre-existing infection at block site.
* Coagulopathy (defined as INR >1.5, Platelets <100,000).
* Known allergy to local anesthetics.
* History of complications from regional anesthesia.
* Emergency or bilateral hernia repair.
* Neurodevelopmental disorders (e.g., cerebral palsy, spina bifida).

Ages: 1 Year to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Estimated)
Dates: Start 2025-11-25 (Estimated); Primary Completion 2026-05-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Time to the first request for rescue analgesia | 24 hours post-operatively
  the interval between the end of surgery (extubation) and the first need for analgesia (paracetamol)

SECONDARY OUTCOMES:
Total intraoperative fentanyl consumption | from the start of general anesthesia until the extubation
Postoperative FLACC (Face, Legs, Activity, Cry, Consolability) pain scores | 24 hours postoperatively
  Each of the five behaviors will be scored on a scale of 0 to 2. The scores are then added together to get a total score, which can range from 0 (no pain) to 10 (severe pain).
Total paracetamol dose in 24 hours | 24 hours postoperatively
Parental satisfaction score | 24 hours postoperatively
  Will be measured using a 5-point Likert scale:
  1. = Extremely dissatisfied
  2. = Unsatisfied
  3. = Neutral
  4. = Satisfied
  5. = Extremely satisfied